CLINICAL TRIAL: NCT04571684
Title: Evaluating the HITSystem to Improve PMTCT Retention and Maternal Viral Suppression in Kenya
Brief Title: Evaluating HITSystem 2.1 to Improve Viral Suppression in Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Kenya Medical Research Institute (Other); Children's Mercy Hospital Kansas City (Other); Global Health Innovations Foundation - Kenya (Unknown); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01MH121245 (NIH); R01MH121245 (NIH)
Record Dates: First submitted 2020-09-22; First posted 2020-10-01 (Actual); Results first posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: HIV; Pregnancy
Keywords: Prevention of mother-to-child transmission (PMTCT) services; maternal viral load monitoring; early infant diagnosis (EID); Kenya; perinatal HIV transmission

STUDY DESIGN:
Intervention Model Description: Matched, cluster randomized controlled design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (HITSystem 2.1) (Experimental): Participants enrolled at intervention sites will received HITSystem 2.1-supported PMTCT services through 6 months postpartum. Interventions received will include: text messages to patients to support medication adherence, appointment attendance, and hospital delivery and algorithm-driven alerts to notify providers when follow up services are missed.
  Interventions: Other: HITSystem 2.1
- Control Arm (Standard of care) (No Intervention): Participants enrolled at control sites will receive standard of care PMTCT services, with no HITSystem 2.1 tracking or follow up.

INTERVENTIONS:
Other: HITSystem 2.1 — HITSystem 2.1 is an intervention that tracks HIV+ pregnant women and their infants to improve the completeness and efficiency of PMTCT services. Key intervention features include: (1) SMS messages sent to enrolled women and mothers to support essential PMTCT services, (2) automated, algorithm-driven alerts for providers when per-guidelines PMTCT services are missed, and (3) automatic enrollment of infants into early infant diagnosis (EID) and linkage with maternal PMTCT file at documentation of infant birth to improve the continuum of care for HIV+ mothers and HIV-exposed infants. The HITSystem 2.1 intervention aims to facilitate complete PMTCT retention and viral load (VL) monitoring with prompt clinical action (adherence support, antiretroviral therapy (ART) regimen change) in the antenatal, delivery, and 6-month postpartum periods to increase viral suppression during windows critical for HIV prevention.
  Arms: Intervention Arm (HITSystem 2.1)

SUMMARY:
The goal of this project is to rigorously evaluate the efficacy of HIV Infant Tracking System 2.1 (HITSystem, an eHealth intervention that uses short message service (SMS) texts to patients and algorithm-driven electronic alerts for providers) to increase retention in guideline-adherent prevention of mother-to-child transmission of HIV services (PMTCT) and to increase viral suppression and appropriate clinical action through the extended period of 6 months postpartum, compared to standard of care PMTCT services in a matched, cluster randomized controlled trial.

DETAILED DESCRIPTION:
Despite progress in providing comprehensive prevention of mother-to-child transmission of HIV (PMTCT) services, significant gaps in the timely uptake and provision of guideline-adherent services and maternal retention in care remain. Such gaps create missed opportunities for preventing mother-to-child transmission and result in nearly 6,100 infants becoming infected with HIV each year in Kenya. Effective interventions that routinize the delivery of evidence-based PMTCT services and foster consistent patient engagement are essential to close the remaining gaps and eliminate mother-to-child transmission of HIV. Building off of a successful R34 grant to develop and pilot test the HITSystem 2.0, an eHealth intervention targeting PMTCT services, the overall goal of this proposal is to use a cluster randomized control design at 12 Kenyan government hospitals to evaluate a modified HITSystem 2.1 intervention. HITSystem 2.1 reflects the 2018 Kenyan PMTCT guidelines, including routine viral load monitoring and interventions to suppress maternal viral load. The investigators aim to evaluate the impact of HITSystem 2.1 to optimize the provision of guideline-adherent services and viral suppression through the antenatal, delivery, and early postpartum periods. Aim 1 of the proposed study will assess the efficacy of the HITSystem 2.1 to increase the proportion of mothers who receive complete PMTCT services (including appointment attendance, medication adherence support, viral load testing, hospital-based delivery, and infant testing per Kenyan National Guidelines) through 6 months postpartum. The investigators hypothesize that mothers receiving the HITSystem 2.1 intervention will have a significantly higher completion rate for guideline-adherence PMTCT services compared to mothers receiving standard of care PMTCT services. In Aim 1b, the investigators will evaluate HITSystem 2.1 implementation using the RE-AIM model to inform sustainable scale up. Aim 2 will assess the efficacy of HITSystem 2.1 to increase viral suppression (<1,000 copies/mL) among pregnant and postpartum women, including those who disengage from care. The investigators hypothesize that mothers at HITSystem 2.1 sites will have higher rates of viral suppression at delivery and 6 months postpartum. Aim 3 will evaluate the cost-effectiveness of the HITSystem 2.1. Driven by differences in PMTCT retention, viral suppression, and modeled estimates of pediatric HIV infections averted, the investigators hypothesize that the HITSystem 2.1 will be cost-effective, based on World Health Organization criteria. This proposal is aimed at improving the quality of PMTCT services in the health facility setting. If efficacious and cost-effective, HITSystem 2.1 holds strong promise for national dissemination.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women living with HIV who present for care at one of the study hospitals by 36 weeks gestation and provide written informed consent are eligible for enrollment in the study.

Exclusion Criteria:

* Pregnant women living with HIV will be excluded from study participation if she has any condition (including drug abuse, alcohol abuse, or psychiatric disorder) that study or hospital staff feel precludes her from providing informed consent.
* Women who transfer care from one study site to another during their PMTCT services will be ineligible for enrollment at their new facility.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1639 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Finocchario-Kessler, PhD, MPH, Principal Investigator — University of Kansas Medical Center
Locations (12):
- Kenya (12):
  - Mariakani Subcounty Hospital, Mariakani, Kilifi County
  - Mtwapa Subcounty Hospital, Mtwapa, Kilifi County
  - Vipingo Subcounty Hospital, Vipingo, Kilifi County
  - Likoni Subcounty Hospital, Likoni, Mombasa County
  - Ambira Subcounty Hospital, Ambira, Siaya County
  - Bondo Subcounty Hospital, Bondo, Siaya County
  - Malanga Subcounty Hospital, Malanga, Siaya County
  - Sigomere Health Center, Sigomere, Siaya County
  - Ukwala Subcounty Hospital, Ukwala, Siaya County
  - Yala Subcounty Hospital, Yala, Siaya County
  - Akala Subcounty Hospital, Siaya
  - Siaya County Hospital, Siaya

IPD SHARING:
Plan to Share IPD: Yes
The investigators will make data collected for aims 1 & 2 available only upon request from users who can show proof of human subject's training and only under a data-sharing agreement that provides for: (1) use of the data only for research purposes, (2) exclusion of any identifying or potentially identifying information in shared analyses, publications, reports, etc., (3) appropriate storage and securing of the data to prevent authorized persons from accessing it, (4) a commitment to destroy or return the data after analyses are completed.
  Data from aim 3 includes costing data for PMTCT services. These data will be shared openly at the dissemination meetings planned at the end of the study, which will include county and national health personnel. Furthermore, these data will be placed in a readily accessible public database.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After participant follow up is complete, data is cleaned, and the final data set is locked
Access Criteria: Upon request from users who can show proof of human subject's training and only under a data-sharing agreement

REFERENCES:
- [Derived] Wexler C, Maloba M, Mokua S, Babu S, Maosa N, Staggs V, Goggin K, Acharya H, Hurley EA, Finocchario-Kessler S. Assessing COVID-related concerns and their impact on antenatal and delivery care among pregnant women living with HIV in Kenya: a brief report. BMC Pregnancy Childbirth. 2024 Jan 9;24(1):46. doi: 10.1186/s12884-023-06216-x. PMID 38195390
- [Derived] Mokua S, Maloba M, Wexler C, Goggin K, Staggs V, Mabachi N, Maosa N, Babu S, Hurley E, Finocchario-Kessler S. Evaluating the efficacy of the HITSystem 2.1 to improve PMTCT retention and maternal viral suppression in Kenya: Study protocol of a cluster-randomized trial. PLoS One. 2022 Jul 26;17(7):e0263988. doi: 10.1371/journal.pone.0263988. eCollection 2022. PMID 35881649

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Sites
Period: Overall Study
Arm/Group | Intervention Arm (HITSystem 2.1) | Control Arm (Standard of Care)
Started | 899; 6 Sites | 740; 6 Sites
Completed | 767; 6 Sites | 627; 6 Sites
Not Completed | 132; 0 Sites | 113; 0 Sites

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm (HITSystem 2.1) | Control Arm (Standard of Care) | Total
Number analyzed (Participants) | 767 | 627 | 1394
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.6 (5.8) | 30.4 (6.0) | 30.5 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 767 | 627 | 1394
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Kenya | 767 | 627 | 1394
Gestational week at enrollment [Mean (Standard Deviation); unit: weeks] | 19.1 (7.8) | 19.9 (7.3) | 19.5 (7.6)
Time of antiretroviral treatment (ART) initiation [Count of Participants; unit: Participants]
  During current pregnancy | 162 | 145 | 307
  <5 yrs prior to current pregnancy | 331 | 228 | 559
  >5 years prior to current pregnancy | 274 | 232 | 506
  Missing | 0 | 22 | 22
Education level [Count of Participants; unit: Participants]
  Less than secondary education | 611 | 508 | 1119
  Completed secondary education | 112 | 74 | 186
  Beyond secondary education | 43 | 41 | 84
  Missing | 1 | 4 | 5
HIV disclosure [Count of Participants; unit: Participants]
  No one | 90 | 89 | 179
  Anyone | 676 | 535 | 1211
  Missing | 1 | 3 | 4
Partner living situation [Count of Participants; unit: Participants]
  No current partner | 52 | 58 | 110
  Live separate from partner | 128 | 104 | 232
  Live with current partner | 581 | 459 | 1040
  Missing | 6 | 6 | 12
Past experience with prevention of mother to child transmission(PMTCT)/early infant diagnosis (EID) [Count of Participants; unit: Participants]
  No | 290 | 272 | 562
  Yes | 477 | 355 | 832
Household income [Count of Participants; unit: Participants]
  <750 KSh | 268 | 224 | 492
  >=750 KSH | 336 | 257 | 593
  Missing | 163 | 146 | 309

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Receiving Complete PMTCT
Description: documented receipt of all of the following: maternal ART initiation, antenatal appointment attendance, facility delivery, EID linkage by 7 weeks of age, maternal viral load testing and clinical action per national guidelines through 6 months postpartum (Table 6). Participants who receive all indicated services per guidelines will be coded as 1 or 'yes'. Participants missing > 1 service will be coded as 0 or incomplete PMTCT services.
Time Frame: 7-15 months (PMTCT enrollment date through 6 months postpartum)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm (HITSystem 2.1) | Control Arm (Standard of Care)
Number analyzed (Participants) | 767 | 627
Participants | 60 | 22

2. Primary Outcome: Viral Suppression
Description: Number of clients with a suppressed viral load(<1000 copies/mL) at delivery
Time Frame: 1-9 months
Population: The overall number of participants analyzed include only those who had a documented viral load test at delivery.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm (HITSystem 2.1) | Control Arm (Standard of Care)
Number analyzed (Participants) | 703 | 581
Participants | 655 | 535

3. Secondary Outcome: PMTCT Retention Duration (Weeks)
Description: The number of weeks women were engaged in PMTCT services
Time Frame: 7-15 months (PMTCT enrollment date through 6 months postpartum)
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Intervention Arm (HITSystem 2.1) | Control Arm (Standard of Care)
Number analyzed (Participants) | 767 | 627
weeks | 48.4 (9.6) | 47.2 (8.1)

4. Secondary Outcome: Antenatal Viral Load (VL) Test Coverage
Description: The number of women receiving viral load testing upon enrolling in prevention of mother to child transmission of HIV services (PMTCT).
Time Frame: Within one month of enrollment in PMTCT
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm (HITSystem 2.1) | Control Arm (Standard of Care)
Number analyzed (Participants) | 767 | 627
Participants | 330 | 137

5. Secondary Outcome: Postnatal Viral Load (VL) Test Coverage
Description: The number of women receiving postpartum viral load testing per the Kenyan national guidelines.
Time Frame: Between delivery and 7 months postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm (HITSystem 2.1) | Control Arm (Standard of Care)
Number analyzed (Participants) | 767 | 627
Participants | 518 | 371

6. Secondary Outcome: Viral Load Test Utility
Description: Number of detectable viral load results with clinical action per guidelines, such as: intensified adherence counseling and/or ARV regimen change
Time Frame: PMTCT enrollment date through 6 months postpartum
Population: Viral load test utility was analyzed only among those participants with a detectable viral load result.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm (HITSystem 2.1) | Control Arm (Standard of Care)
Number analyzed (Participants) | 35 | 29
Participants | 28 | 18

7. Secondary Outcome: Turnaround Time of Viral Load Sample Collection to Patient Notification
Description: The median number of days from the date of VL sample collection to patient notification, among all viral load tests
Time Frame: PMTCT enrollment date through 6 months postpartum
Population: Turnaround time was measured among all viral load samples taken in the antenatal and/or postpartum periods.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Intervention Arm (HITSystem 2.1) | Control Arm (Standard of Care)
Number analyzed (Participants) | 767 | 627
days | 35 [21 to 56.5] | 35 [23 to 48.3]

8. Secondary Outcome: Antiretroviral Therapy (ART) Adherence
Description: The number of participants with ART adherence > 95%
Time Frame: 7-15 months (PMTCT enrollment date through 6 months postpartum)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm (HITSystem 2.1) | Control Arm (Standard of Care)
Number analyzed (Participants) | 767 | 627
Participants | 466 | 200

ADVERSE EVENTS:
Time Frame: We collected information on adverse events from the time of participant enrollment through 6 months postpartum, up to a total of 15 months.
Arm/Group | Intervention Arm (HITSystem 2.1) | Control Arm (Standard of Care)
All-Cause Mortality (participants affected / at risk) | 14/899 | 22/740
Serious Adverse Events (participants affected / at risk) | 41/899 | 41/740
Other Adverse Events (participants affected / at risk) | 0/899 | 0/740
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Arm (HITSystem 2.1) (N=899) | Control Arm (Standard of Care) (N=740)
Pregnancy Loss (Pregnancy, puerperium and perinatal conditions) | 41 | 41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-10-03): https://cdn.clinicaltrials.gov/large-docs/84/NCT04571684/Prot_SAP_ICF_000.pdf